CLINICAL TRIAL: NCT02863874
Title: Comparison of VicrylPlus® Versus Vicryl® for Surgical Repair of Perineal Tears; a Prospectively Randomized Controlled Trial
Brief Title: The PLUS Study: Comparison of VicrylPlus® Versus Vicryl® for Repair of Perineal Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015/774
Record Dates: First submitted 2016-04-29; First posted 2016-08-11 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Skin Structures and Soft Tissue Infections; Wound Infection
Keywords: Perineal tear; Labor; Triclosan
MeSH Terms: conditions — Soft Tissue Infections; Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vicryl® (Active Comparator): The vaginal or and perineal tear is sutured continuously with Vicryl®. The instruments for suturing and the bedcover are clean whereas the gloves are sterile.
  Interventions: Device: Vicryl®
- VicrylPlus® (Active Comparator): The vaginal or and perineal tear is sutured continuously with VicrylPlus®. The instruments for suturing and bedcover are clean whereas the gloves are sterile.
  Interventions: Device: VicrylPlus®

INTERVENTIONS:
Device: VicrylPlus® — Suture
  Arms: VicrylPlus®
Device: Vicryl® — Suture
  Arms: Vicryl®

SUMMARY:
INTRODUCTION It is estimated that over 80% of women who give vaginal birth will sustain some form of perineal tear and of these 60-70% will require suturing. It is of great importance that operators are familiar with the best suturing technique and suture material in order to minimize possible associated short- and long-term sequelae. There is evidence for suturing continuously to reduce postoperative pain and superficial dyspareunia, but the choice of suture-material is still debated. The function of a suture is to close the wound to minimize the bleeding, the risk for infection and to adapt the wound edges to promote anatomic correct healing. Infection results in softened wound edges, shirked sutures, pain and dehiscence. Delayed and/or compromised wound healing is correlated with impaired strength in the affected tissue. Reported frequency of infection after first and second degree tear is between 1 and 11% where the discrepancy most likely is due to poor registration and follow-up. In 2004 Polyglactin 910 was launched with a new antibacterial coating of Triclosan (VicrylPlus®). Studies suggest a correlation between the use of VicrylPlus® and a reduction of up to 30% of surgical site infections (SSI) compared to conventional sutures in a non-colonized wound.

OBJEKTIVE: The primary objective is to compare infection rates and pain intensity when using Vicryl® versus VicrylPlus® for perineal repair after delivery. Secondly, to show if there is a difference in sequelae (pelvic floor dysfunction) after one year between the two groups.

METHODS The participants are randomly allocated to continuously suturing with either Vicryl® or VicrylPlus®. Sealed identical-looking envelopes are prepared and placed in the delivery room (randomized into blocks of 50) containing randomization number, sutures, declaration of informed consent and questionnaires. The participants are instructed to fill in the first questionnaire after 7 days and the second questionnaire after 8 weeks post partum. After 8 weeks all participants are offered a routine visit to the "out-patient clinic". After one year an internet-based survey will be sent out to the participants. In case of complains/signs of deficient healing after one year, the woman will be offered a clinical control. Data will be analyzed according to intention to treat and per-protocol".

DETAILED DESCRIPTION:
HYPOTHESIS: VicrylPlus® is superior to Vicryl® in terms of infection rate, delayed perineal wound healing and short-/longterm perineal discomfort.

Methods: Women given birth at Skåne University hospital after November 23, 2015 are assessed for eligibility. The hospital consist of two labor wards with approximately 9.000 deliveries pr year. After birth and in case of a first, second or third degree tear, the "labor-responsible" midwife or doctor prepares the patient for the required suture procedure. The two sutures used in this project are not new to the staff, before the beginning of the study both sutures were available on the delivery rooms and randomly used dependent on the midwife's/doctor's preference. Also, before study-start all midwifes/doctors were carefully instructed in detection and classification of perineal tears and the corresponding suturing technique. There is evidence for suturing deep and long tears in the vagina and tears in perineum continuously why we have educated and trained our staff to suture by this technique (e-learning and practical training). Tears will be sutured mainly by midwives and in case of doctor assistance this will be recorded in the obstetrical chart. The delivery course, degree of laceration, suture-procedure are always documented in our electronic obstetrical record accordingly to predefined standards (Obstetrix, Siemens). If the woman is enrolled in the study the randomization number will be incorporated in the operation description.

After identification of a tear requiring continuously suturing (and not only a few stitches) the personal will kindly ask the woman to participate in the study. The woman will be introduced to the reason for conducting the study and to the questions. If she do not agree or is unable for enrollment, or if the midwife is un-certified in continuously suturing, the midwife can choose the suture she usually prefers.

If the woman agrees, she will be randomly allocated to suturing with either Vicryl® or VicrylPlus®, CT-1, 2/0 gauge by drawing a sealed pre-packed and identical looking envelope whereafter written informed consent will be obtained. The envelope contains the randomization number (randomized into blocks of 50 by Randomization.com), two packets of identical sutures, an envelope to the patient with the questionnaires and a prepaid returning envelope. The type of suture will be blinded for the participants and for possible contacts to medical staff after discharge, but not to the suturing midwife/doctor who is carefully instructed not to disclose the origin of the suture used. If there is need for more than 2 sutures the staff can bring more material from our sterile depot. Randomization number, the woman's personal number and the woman's and the operator's signature are all noted on the written patient consent. The document will be returned to a locked box. Once in a week the responsible investigator (Nana Wiberg) empties the box. The randomization number, date of inclusion, personal number, telephone number will be noted by NW in the specific study protocol to which only Kristine Lund Sønnichsen (KLS) and NW have access. The informed consent will thereafter be placed into a locked cabinet. The patient is instructed to fill in the questionnaire at respectively 7 days and 8 weeks postpartum and in the meantime bring it with her, in case of a clinical control. The questionnaire consists of a general information sheet where the woman fills in information about education, body mass index (BMI), previous and actual pregnancy and deliveries. The other sheet consists of a visual analogue scale (VAS scale), questions about eventually use of painkillers and "signs-of-infection" questions accordingly to the CDC criteria. The third part is only used in case of contact with medical staff after discharge. All non-respondents will be contacted primarily by telephone and secondarily by sending a reminding letter by one of the investigators (KLS or NW) if the questionnaire is not received within a week after expected deadline (calculated from date of inclusion). When the questionnaire is received the answers are noticed together with the obstetrical data of interest in the study protocol by one of the investigators (KLS). All obstetrical data are extracted from the same database (Obstetrix). After one year the patient will be asked to fill in an electronic internet based survey and in case of complains/symptoms of deficient healing the woman will be invited to a clinical control.

Statistics Calculation The sample size to detect a 50% reduction in infections from an estimated prevalence of 10% gives 474 participants in each arm to detect this difference with 80% power at 5% significance level, two tailed. Data will be analyzed according to intention to treat and per-protocol. Continuous variables will be presented as mean ± standard deviation, median, range and categorical variables as number (percentage). For comparison between groups following test will be used; the unpaired t-test for continuous normally distributed data, the Mann-Whitney U-test for continuous skew distributed data and the χ2 test for categorical variables. Frequency data will be presented as odds ratios with 95% confidence interval. Spearman's rank correlation will be used to analyze correlations between continuous variables. P < 0.05 is considered statistically significant. The IBM Statistical Package for Social Sciences, Windows version 22 will be used (SPSS, Inc., Chicago, IL, USA) for statistical analysis. The CONSORT 2010 Statement will be met. An independent steering committee will conduct interim analysis after 800 inclusions to estimate when to close the study. Women in need of continuously suturing but not included in the study are noticed in the protocol. Women included but not answering the questionnaire is considered to be a part of the trial. A flow chart will be used to visualize the study group/exclusions and dropouts.

Ethical aspects The study is approved by the local ethical board, Lund, Sweden (Dnr 2015/10).

Sideeffects There is no reason to believe that this study will inflict any harm or any other side effects to the participants or the operator. Triclosan is approved by FDA (U.S. Food and Drug Administration) and there are no reports or evidence for any side effects including allergic reactions or induction of antibiotic resistance.

ELIGIBILITY:
Inclusion

* Vaginal delivery complicated by a spontaneously first, second or third degree tear with need of continuously suturing
* Woman with episiotomy
* Able to read and understand Swedish

Exclusion

* Previously perineal surgery other than primary repair after delivery
* Birth of a stillborn infant
* HIV or active Hepatitis B/C infection
* Severe perineal warts or varicose veins
* The operator is uncomfortable with continuous suturing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1890 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Incidence of wound infection in vaginal and perineal tears after suturing with normal braided suture (Vicryl®) versus antibacterial braided suture (VicrylPlus®). | 4 weeks
  Presence of infection determined by a certified physician according to CDC's Criteria for Defining a Surgical Site Infection.

SECONDARY OUTCOMES:
Difference in self-reported pain after suturing vaginal and perineal tears with normal braided or antibacterial braided suture. | 8 weeks
  The woman is instructed to fill in the VAS scale (visual analog scale)
Number of patients who need or are resutured within one year after delivery for each suture | one year after delivery
  From EMR these data will be retrieved
Number of patients with superficial/deep dyspareunia or pelvic floor dysfunction one year after delivery for each suture | one year after delivery
  The participants will be asked to fill in a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nana Wiberg, MD, PhD, Principal Investigator — Senior consultant, Dept of Gyn et Obst, SUS, Lund, Sweden.
Locations (1):
- Department of Gynecology and Obstetrics, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang ZX, Jiang CP, Cao Y, Ding YT. Systematic review and meta-analysis of triclosan-coated sutures for the prevention of surgical-site infection. Br J Surg. 2013 Mar;100(4):465-73. doi: 10.1002/bjs.9062. Epub 2013 Jan 21. PMID 23338685
- [Background] McCandlish R, Bowler U, van Asten H, Berridge G, Winter C, Sames L, Garcia J, Renfrew M, Elbourne D. A randomised controlled trial of care of the perineum during second stage of normal labour. Br J Obstet Gynaecol. 1998 Dec;105(12):1262-72. doi: 10.1111/j.1471-0528.1998.tb10004.x. PMID 9883917
- [Background] Kettle C, Hills RK, Jones P, Darby L, Gray R, Johanson R. Continuous versus interrupted perineal repair with standard or rapidly absorbed sutures after spontaneous vaginal birth: a randomised controlled trial. Lancet. 2002 Jun 29;359(9325):2217-23. doi: 10.1016/S0140-6736(02)09312-1. PMID 12103284
- [Background] Kettle C, Dowswell T, Ismail KM. Absorbable suture materials for primary repair of episiotomy and second degree tears. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD000006. doi: 10.1002/14651858.CD000006.pub2. PMID 20556745
- [Background] Johnson A, Thakar R, Sultan AH. Obstetric perineal wound infection: is there underreporting? Br J Nurs. 2012 Mar 8-21;21(5):S28, S30, S32-5. doi: 10.12968/bjon.2012.21.Sup5.S28. PMID 22489339
- [Background] Gartti-Jardim EC, de Souza AP, Carvalho AC, Pereira CC, Okamoto R, Magro Filho O. Comparative study of the healing process when using Vicryl(R), Vicryl Rapid(R), Vicryl Plus(R), and Monocryl(R) sutures in the rat dermal tissue. Oral Maxillofac Surg. 2013 Dec;17(4):293-8. doi: 10.1007/s10006-012-0380-3. Epub 2012 Dec 28. PMID 23269361
- [Background] Ford HR, Jones P, Gaines B, Reblock K, Simpkins DL. Intraoperative handling and wound healing: controlled clinical trial comparing coated VICRYL plus antibacterial suture (coated polyglactin 910 suture with triclosan) with coated VICRYL suture (coated polyglactin 910 suture). Surg Infect (Larchmt). 2005 Fall;6(3):313-21. doi: 10.1089/sur.2005.6.313. PMID 16201941
- [Background] Edmiston CE, Seabrook GR, Goheen MP, Krepel CJ, Johnson CP, Lewis BD, Brown KR, Towne JB. Bacterial adherence to surgical sutures: can antibacterial-coated sutures reduce the risk of microbial contamination? J Am Coll Surg. 2006 Oct;203(4):481-9. doi: 10.1016/j.jamcollsurg.2006.06.026. Epub 2006 Aug 22. PMID 17000391
- [Background] Fernando R, Sultan AH, Kettle C, Thakar R, Radley S. Methods of repair for obstetric anal sphincter injury. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD002866. doi: 10.1002/14651858.CD002866.pub2. PMID 16855993
- [Background] Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. Am J Infect Control. 2008 Jun;36(5):309-32. doi: 10.1016/j.ajic.2008.03.002. No abstract available. PMID 18538699
- [Derived] Sonnichsen K, Isberg PE, Elers J, Zaigham M, Wiberg N. The PLUS study: efficacy of triclosan coated suture (VicrylPlus(R)) to reduce infection in primary suture of childbirth related perineal tears - a randomized controlled trial. Matern Health Neonatol Perinatol. 2025 May 5;11(1):13. doi: 10.1186/s40748-025-00211-0. PMID 40320545